CLINICAL TRIAL: NCT00832078
Title: Test Catheter Pilot Study in Healthy Volunteers
Acronym: Test catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DK058CC
Record Dates: First submitted 2009-01-26; First posted 2009-01-29 (Estimated); Results first posted 2012-09-05 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Other): SCCM (SpeediCath Compact Male catheter) then SC (SpeediCath cathter) on test day 1. SC then SCCM on test day 2
  Interventions: Device: SpeediCath Compact Male; Device: Speedicath
- Group B (Other): SC (SpeediCath cathter)then SCCM (SpeediCath Compact Male catheter) on test day 1. SCCM then SC on test day 2
  Interventions: Device: SpeediCath Compact Male; Device: Speedicath

INTERVENTIONS:
Device: SpeediCath Compact Male — CH 12 hydrophilic coated intermitten compact catheter
Device: Speedicath — CH 12 hydrophilic coated intermittent coated catheter

SUMMARY:
The purpose of this study is to evaluate the safety of an intermittent catheter in comparison with an already existing catheter on the market. The study is a randomised, single blinded, cross-over study including 25 healthy males.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Male
* Signed informed consent
* Negative urine multistix

Exclusion Criteria:

* Abnormalities, diseases or surgical procedures performed in the lower urinary tract

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2009-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshopsitalet, Copenhagen, København Ø, Denmark

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 28 participants enrolled in study. 2 were excluded before randomization as they did not comply with inclusion criteria. One was excluded from study (ITT) as participants dropped out before having any data recorded.
Groups:
- Group A: Test day 1: first SCCM then SC; Test day 2: first SC then SCCM; this gives 4 catherizations per participant
- Group B: Test day 1 first SC then SCCM; Test day 2 first SCCM then SC; this gives 4 catherizations per participant
Period: Test Day 1- 1 Period
Arm/Group | Group A | Group B
Started | 13 | 12
Completed | 13 | 12
Not Completed | 0 | 0
Period: Test Day 1-2 Period
Arm/Group | Group A | Group B
Started | 13 | 12
Completed | 13 | 10
Not Completed | 0 | 2
Not completed — Lack of Efficacy | 0 | 2
Period: Test Day 2 - 1 Period
Arm/Group | Group A | Group B
Started | 13 | 10
Completed | 13 | 10
Not Completed | 0 | 0
Period: Test Day 2 - 2 Period
Arm/Group | Group A | Group B
Started | 13 | 10
Completed | 12 | 10
Not Completed | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 27.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 25
Region of Enrollment [Number; unit: participants]
  Denmark | 25

OUTCOME MEASURES:

1. Primary Outcome: Discomfort
Description: Discomfort measured on a Visual Analog Scale (VAS) from 0 (no discomfort) to 10 (worst imaginable discomfort)
Time Frame: After each catheterisation
Population: The number analized was the number of participants catherised with each catheter at least onze during the study(SC or SCCM)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Test Catheter SCCM: The Test catheter SpeediCath Compact Male (SCCM)
- Standard Catheter SC: The Stanard catheter SpeediCath (SC)
Arm/Group | Test Catheter SCCM | Standard Catheter SC
Number analyzed (Participants) | 23 | 25
units on a scale | 2.25 (1.5) | 2.52 (1.8)

2. Secondary Outcome: Handling
Time Frame: After each catheterisation
Reporting Status: Not Posted

3. Secondary Outcome: Preference
Time Frame: At study termination
Reporting Status: Not Posted

4. Secondary Outcome: Haematuria
Time Frame: After each catheterisation
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Test Catheter | Standard Catheter
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less